CLINICAL TRIAL: NCT02718781
Title: Community Health Campaign: Fitter Families Project
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Hong Kong (Other)
Responsible Party: Principal Investigator, Dr. Steven C. Shen, Post-doctoral Fellow, The University of Hong Kong
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: UW15-401
Record Dates: First submitted 2016-03-10; First posted 2016-03-24 (Estimated); Last update posted 2017-07-05 (Actual); Status verified 2017-07

CONDITIONS: Health Behavior
MeSH Terms: conditions — Health Behavior

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Talk and leaders (Experimental): This group will comprise of health talk and regular contact with community leaders.
  Interventions: Behavioral: Health talk; Behavioral: Regular contact with community leaders
- Talk, leaders and equipment (Experimental): This group will comprise of health talk and regular contact with community leaders. Moreover, a home-based equipment (handgrip) will be delivered to them
  Interventions: Behavioral: Health talk; Behavioral: Regular contact with community leaders; Device: Handgrip
- Talk (Active Comparator): This group will comprise of a health talk only.
  Interventions: Behavioral: Health talk

INTERVENTIONS:
Behavioral: Health talk — Health talk on zero-time exercise.
Behavioral: Regular contact with community leaders — Regular contact with community leaders to remind them do zero-time exercise.
  Arms: Talk and leaders; Talk, leaders and equipment
Device: Handgrip — This is a home-based equipment
  Arms: Talk, leaders and equipment

SUMMARY:
In recent years, Hong Kong has been undergoing rapid changes with macro social and economic trends. The increasingly complex and diverse family structure contribute to concerns regarding the well-being of families in Hong Kong, including their health, happiness and harmony (FAMILY 3Hs). Family life and health education should be strengthened to meet the increasing needs of promoting healthy active lifestyle among Hong Kong families. In this connection, the FAMILY Project initiates the Fitter Families Project (FFP) with a focus on "FAMILY Holistic Health", will be conducted in order to increase the awareness of the importance of FAMILY 3Hs. FFP is a community-based research project with 3 main components - train-the-trainers programs, community-based family interventions and public education events. It is expected that trainees from the train-the-trainers programs will acquire adequate skills to organize community-based health education programs effectively. Participants of the community-based family interventions will gain knowledge on family holistic health and live a healthy active lifestyle. Attendees of the public education events will become more aware of the importance of FAMILY 3Hs.

DETAILED DESCRIPTION:
In 2011, United Nations (UN) addressed the prevention and control of four non-communicable diseases (NCDs: cancer, cardiovascular disease, chronic respiratory disease, and diabetes mellitus) worldwide. The UN, in its Political Declaration, recognized the critical importance of reducing the exposure to the common modifiable risk factors for NCDs, namely, tobacco use, unhealthy diet, physical inactivity, and the harmful use of alcohol. In Hong Kong, NCDs are responsible for more than 85% of all deaths and most of these are preventable. FAMILY Project Cohort Study (2014) also found that 88.6% of Hong Kong people had inadequate vegetable and fruit intake, 70.6% had inadequate physical exercise, 26.4% were overweight and 5.4% were obese. Hong Kong, being the most westernized and developed city of China, can take a leading role in promoting and implementing the UN Political Declaration.

Families worldwide have been undergoing rapid changes with macro, social and economic trends. Demographic shifts, economic upheavals, changing societal norms and values, immigration across national borders and migration within nations are creating new and altered structures, processes and relationships within families. The increasingly complex and diverse family structure contributes to concerns regarding the well-being of families in Hong Kong, including their health, happiness and harmony (FAMILY 3Hs). Family life and health education should be strengthened to meet the increasing needs of promoting healthy lifestyle among Hong Kong families. The results from the baseline findings of FAMILY Project Cohort Study (2014) revealed that only 27.9% of the participants considered themselves to be 'happy', while 15.6% of the participants were classified as 'unhappy'. Nearly one-third (30.7%) of the participants reported having experienced at least one stressful life event in the previous year due to heavier workload (10.8%), serious health problems of a family member (6.8%), worsening financial situation (6.2%), health problems of oneself (5.1%), or death of a family member (4.7%). Furthermore, more than half of the participants (52.5%) reported having some source of dyadic conflicts with family members. In response to these changes in the contexts and nature of the family, the Fitter Families Project (FFP) with a focus on "FAMILY Holistic Health", will be conducted in order to increase the awareness of the importance of FAMILY 3Hs.

There are several definitions of family health. On the functional level, the terms family health, family functioning, and healthy family are often used interchangeably. Family health has been described as complex system, interactions, relationships and processes with the potential to enhance both well-being and the entire household's health, and routines in the family may affect family health. Despite the different perspectives in the definitions, family health should be holistically defined, encompass both wellness and illness variables and focus on the interactive, developmental, functional, psychosocial, and health processes of family experience. Therefore, family health may be described as a dynamic process that maintains or changes the relative state of well-being, including elements of family systems, such as biological, psychological, spiritual, and sociocultural aspects. Hence, the FFP focuses on "FAMILY Holistic Health" which is to emphasize a more comprehensive and wide reaching aim and includes physical, mental and social health and well-being.

Over the past six years, the FAMILY project has been working on community-based projects to promote FAMILY 3Hs. Since 2010, the Christian Family Service Centre (CFSC) in collaboration with the School of Public Health of the University of the Hong Kong (HKU) implemented a community-based Learning Families Project (LFP) to promote family health, happiness and harmony (3Hs). As a component of the FAMILY Project, the LFP had built up an effective practice model through collaboration among various project partners and showed good evidence of effectiveness in developing a learning culture in the families, enhancing family communication time and quality, increasing neighborhood cohesion and resilience and promoting FAMILY 3Hs. Therefore, the FFP is developed based on the strong foundation of the LFP in the previous years. In view of the health challenges locally and globally, the new phase of FAMILY project will put more emphasis on health in the upcoming three years. Following the theme on FAMILY 3Hs, the FFP focuses on family holistic health with emphasis on the interaction and integration of both physical and psychosocial health.

In Hong Kong, most 'health projects' only focus on individual's physical health and usually separate physical from mental or psychosocial health. This new project focuses not only on individuals' health but on the whole family and holistic health. The investigators strive to help family members influence each other to have better holistic health. The focus on family is a new and unique concept which is an innovative, long-term and highly sustainable approach at the community level. With the involvement of family members, Hong Kong families can develop and change their lifestyles which impact on families' health. The investigators will use a family-focused approach and adopt a holistic perspective to design a sustainable family holistic health intervention model in the community to meet the global health challenges identified by UN.

The innovative family holistic health intervention model will emphasize on the interaction and integration of physical health and psychosocial health, using physical exercise as the platform to promote fitter families, which will ultimately enhance the FAMILY 3Hs. Thus, the ultimate objective of this community-based project is "FAMILY holistic health" for FAMILY 3Hs.

In practice, the investigators will use innovative integrated public health theories and minimal methods to plan brief, simple and cost-effective interventions targeted at families, with collaboration with experienced NGO partners and community stakeholders. Hence, a larger number of people will be able to benefit from the program, leading to greater sustainability and wider dissemination as the administration of project will be easier and the costs will be lower. The "FAMILY Holistic Health" community-based project aims at promoting a higher level of physical exercise for people of all ages which will enhance family interaction, pleasure and well-being. The project can help families to build positive attitudes with stronger motivation for family members to improve their holistic health by encouraging each other to have healthy active lifestyle and enjoy the processes with quick and measurable benefits.

The evaluations conducted will be vigorous and evidence generating with quantitative and qualitative methods and follow-ups to assess behavioral changes and improvements in the key components of family well-being. The data will be provided to the participants for developing their own health action plan. In order to assess the effectiveness of the interventions on improving individual and family well-being and for future program development, the data will also be used for program evaluation. Thus, this proposal is to seek approval from IRB to collect data from the participants, to use the data for in depth analyses, and to write up scientific papers based on the findings.

ELIGIBILITY:
Inclusion Criteria:

* Cantonese speaking, Intact verbal and hearing abilities for interpersonal communication, Reading and writing abilities for questionnaire completion, aged 12 or above

Exclusion Criteria:

* Participants who fail to meet the inclusion criteria

Min Age: 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 953 (Actual)
Dates: Start 2015-09 (Actual); Primary Completion 2016-12 (Actual); Study Completion 2017-06 (Actual)

PRIMARY OUTCOMES:
Changes in family harmony from baseline to 3 months after intervention | Baseline, at 1 month after intervention, and at 3 months after intervention
  Family harmony will be assessed by a 0-10 score at 3 time points
Changes in family happiness from baseline to 3 months after intervention | Baseline, at 1 month after intervention, and at 3 months after intervention
  Family happiness will be assessed by a 0-10 score at 3 time points
Changes in family health from baseline to 3 months after intervention | Baseline, at 1 month follow-up, and at 3 months after intervention
  Family health will be assessed by a 0-10 score at 3 time points

SECONDARY OUTCOMES:
Changes in knowledge on zero-time exercise from baseline to 3 months after intervention | Baseline, immediately after intervention, at 1 month after intervention, and at 3 months after intervention
  Questionnaire will be used to investigate the changes in participants' knowledge on zero-time exercise.
Changes in attitude towards performing zero-time exercise from baseline to 3 months after intervention | Baseline, immediately after intervention, at 1 month after intervention, and at 3 months after intervention
  Questionnaire will be used to investigate the changes in participants' attitude towards performing zero-time exercise.
Changes in intention at performing zero-time exercise from baseline to 3 months after intervention | Baseline, immediately after intervention, at 1 month after intervention, and at 3 months after intervention
  Questionnaire will be used to investigate the changes in participants' intention at performing zero-time exercise.
Changes in the frequency and amount on performing exercise from baseline to 3 months after intervention | Baseline, at 1 month after intervention, and at 3 months after intervention
  Questionnaire will be used to investigate the changes in participants' frequency and amount on performing moderate exercise (e.g. cycling or quick walking), vigorous exercise (e.g. swimming or jogging), zero-time exercise and walking.
Changes in neighborhood cohesion from baseline to 3 months after intervention | Baseline, at 1 month after intervention, and at 3 months after intervention
  Questionnaire will be used to investigate the changes in participants' neighborhood cohesion by a 5-items scale.
Changes in utilization of community resources from baseline to 3 months after intervention | Baseline, at 1 month after intervention, and at 3 months after intervention
  Questionnaire will be used to investigate the changes in participants' utilization of community resources to perform exercise.
Changes in grip strength (kg) from baseline to 3 months after intervention | Baseline, at 1 month after intervention, and at 3 months after intervention
  Grip strength will be assessed by a hand grip strength measurement instrument.
Changes in chair stand (times) from baseline to 3 months after intervention | Baseline, at 1 month after intervention, and at 3 months after intervention
  Chair stand will be assessed by a test counting times of chair stand in 30 seconds.
Changes in single leg stand (s) from baseline to 3 months after intervention | Baseline, at 1 month after intervention, and at 3 months after intervention
  Single leg stand will be assessed by a test measuring the longest duration of single leg stand in 120 seconds.
Changes in seat and reach (cm) from baseline to 3 months after intervention | Baseline, at 1 month after intervention, and at 3 months after intervention
  Seat and reach will be assessed by a ruler.
Changes in body fat (%) from baseline to 3 months after intervention | Baseline, at 1 month after intervention, and at 3 months after intervention
  Changes in body fat will be assessed by a standard body fat measuring scale.
Changes in body weight (kg) from baseline to 3 months after intervention | Baseline, at 1 month after intervention, and at 3 months after intervention
  Changes in body weight will be assessed by a standard body fat measuring scale.
Satisfaction towards the program | Immediately after intervention
  Questionnaire will be used to investigate the participants' satisfaction towards the program immediately after intervention.

CONTACTS AND LOCATIONS:
Overall Officials: Chen Shen, PhD, Principal Investigator — The University of Hong Kong
Locations (1):
- Christian Family Service Center, Hong Kong, Hong Kong

REFERENCES:
- [Background] Anderson KH, Tomlinson PS. The family health system as an emerging paradigmatic view for nursing. Image J Nurs Sch. 1992 Spring;24(1):57-63. doi: 10.1111/j.1547-5069.1992.tb00700.x. PMID 1541473
- [Background] Denham SA. Family routines: a structural perspective for viewing family health. ANS Adv Nurs Sci. 2002 Jun;24(4):60-74. doi: 10.1097/00012272-200206000-00010. PMID 12699277
- [Background] Leung GM, Ni MY, Wong PT, Lee PH, Chan BH, Stewart SM, Schooling CM, Johnston JM, Lam WW, Chan SS, McDowell I, Lam TH, Pang H, Fielding R. Cohort Profile: FAMILY Cohort. Int J Epidemiol. 2017 Apr 1;46(2):e1. doi: 10.1093/ije/dyu257. PMID 25617647
- [Background] Wacharasin C, Theinpichet S. Family nursing practice, education, and research: what is happening in Thailand? J Fam Nurs. 2008 Nov;14(4):429-35. doi: 10.1177/1074840708327515. PMID 19139157
- [Background] Yoshikawa H. Integrating methods in the science of family health: new directions from an institute of medicine workshop report. Arch Pediatr Adolesc Med. 2012 Jul 1;166(7):659-61. doi: 10.1001/archpediatrics.2012.510. No abstract available. PMID 22751883
- See also: United Nations. (2011). Political declaration of the high-level meeting of the general assembly on the prevention and control of non-communicable diseases. — http://ncdalliance.org/sites/default/files/rfiles/UN%20HLM%20Political%20Declaration%20English.pdf